CLINICAL TRIAL: NCT05402540
Title: Effectiveness of Strain Counter Strain Technique Verses Active Release Technique in Adhesive Capsulitis
Brief Title: Effectiveness of SCS Technique Verses ART in Adhesive Capsulitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/01206 Khizar Hayat
Record Dates: First submitted 2022-04-21; First posted 2022-06-02 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Adhesive Capsulitis
Keywords: ADHESIVE CAPSULITIS; SHOULDER PAIN; Range of Motion; Shoulder Muscle Strength
MeSH Terms: conditions — Bursitis; Shoulder Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- STRAIN COUNTER STRAIN GROUP (Experimental): Strain Counter Strain Technique in combination with conventional physiotherapy
  Interventions: Other: STRAIN COUNTER STRAIN GROUP
- ACTIVE RELEASE TECHNIQUE GROUP (Experimental): Active Release Technique in combination with conventional physiotherapy
  Interventions: Other: ACTIVE RELESAE TECHNIQUE GROUP

INTERVENTIONS:
Other: STRAIN COUNTER STRAIN GROUP — Strain Counterstrain Technique in combination with conventional physiotherapy (Hot pack, Codman"s exercises, active assisted exercises, Pendulum exercises, Finger Ladder Exercise, Maitland mobilization of shoulder joint.
  Therapist palpate surrounding and opposing tissues to locate trigger point by using one or two finger pads to monitor fasciculation and MTrP.
  Hold the POC (position of comfort) until fasciculation decreases significantly or ceases. Average positions hold time while pressure is 90 s to 3 min.
  Release tissue or joint slowly and reassess. Each patient will receive total 6 sessions (3sessions/week) over a period of 2 weeks.
  Assessment would be done on baseline and after every three sessions.
  Arms: STRAIN COUNTER STRAIN GROUP
Other: ACTIVE RELESAE TECHNIQUE GROUP — Active Release Technique in combination with conventional physiotherapy (Hot pack, Codman"s exercises, active assisted exercises, Pendulum exercises, Finger Ladder Exercise, Maitland mobilization of shoulder joint.
  The targeted muscle will be palpated while the therapist will looks for localized tenderness or trigger points with referred pain elicitation.
  With the thumb therapist will relieve the trigger point. In ART the particular muscle is taken from shortened to lengthened position or from lengthened to shortened position.
  Duration of treatment will be 8-15 minutes. Each patient will receive total 6 sessions (3sessions/week) over a period of 2 weeks.
  Assessment would be done on baseline and after every three sessions.
  Arms: ACTIVE RELEASE TECHNIQUE GROUP

SUMMARY:
To find out the effectiveness of Strain Counter strain Technique verses Active Release Technique on upper trapezius, subscapularis, anterior fiber of deltoid and supraspinatus muscles trigger points in adhesive capsulitis in term of pain intensity, range of motion and muscle strength.

DETAILED DESCRIPTION:
Frozen shoulder, also known as adhesive capsulitis, is defined as "a condition of uncertain aetiology, characterized by significant restriction of both active and passive shoulder motion that occurs in the absence of a known intrinsic shoulder disorder". Prevalence ranges from 2% to 5% in general population. It is relatively more common in women than men, often in non-dominant arm and age between 40 and 60 years. Frozen shoulder was also termed as adhesive capsulitis (AC) due to its chronic inflammatory process. Painful stiffness of the shoulder can adversely affect activities of daily living and consequently impair quality of life. Adhesive capsulitis can be primary or secondary. Primary (or idiopathic) adhesive capsulitis can occur spontaneously without any specific trauma or inciting event. Secondary adhesive capsulitis is often observed after periarticular fracture dislocation of the glenohumeral joint or other severe articular trauma.

Dr. Lawrence Jones, an osteopathic physician, is credited with the discovery of the therapy; he initially called it Positional release technique (PRT) and later coined the term strain counterstrain. Originally termed strain-counterstrain, is a therapeutic technique that uses trigger points (TrPs) and a position of comfort (POC) to resolve the associated dysfunction. A gentle and passive technique, SCS has been advocated for the treatment of acute, subacute and chronic dysfunction in people of all ages.A number of studies have reported the use of strain/counterstrain in combination with other interventions for treating a variety of disorders, including chondromalacia patellae, low back pain, and cervicothoracic pain.

Active Release Techniques (ART) is a soft tissue method that focuses on relieving tissue tension via the removal of fibrosis/adhesions which can develop in tissues as a result of overload due to repetitive use. The goals of ART are to restore optimal tissue texture, tension and movement, restore the strength, flexibility, function, and relative translation between soft tissue layers, release any soft tissue restrictions, entrapped nerve, restricted circulatory structures, or lymphatic restrictions. ART is used to find the specific tissues that are restricted, physically work on the soft tissues back to their normal texture, tension, and length by using various hand positions and soft tissue manipulation methods.

Active release technique and capsular stretch with conventional therapy is more effective in increasing ROM and decreasing pain of frozen shoulder rather alone capsular stretch with conventional therapy. These changes are clinically significant. Both positional release and muscle energy techniques were shown to be effective in improving functional ability of shoulder in Adhesive Capsulitis, but muscle energy technique was better than positional release technique..Both ART and SCS technique play important role in decreasing hamstring tightness but Active Release Technique is more effective physiotherapeutic intervention than strain counterstrain technique in reducing hamstrings tightness instantly.

Active Release Techniqueand Strain Counterstrain have been proved to be effective in many conditions like low back pain, chronic neck pain, tennis elbow, CTS and shoulder pain. ART and SCS has also been proved effective in treating upper trapezius, subscapularis SCM, hamstring muscle trigger point in comparison with other treatment protocol. But there is limited studies done on comparing these two techniques i.e ART and SCS for the adhesive capsulitis and specifically the use of ART and SCS for AC induced trigger points in different muscles of shoulder. Hence, the aim of present study is to compare the effectiveness of Active release technique and Strain counterstrain technique in adhesive capsulitis induce trigger points in different shoulder muscle in term of pain, ROM and muscle strength.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic Adhesive Capsulitis (AC)
* Stage 2 AC
* Both genders
* ROM limitation in capsular pattern
* AC having myofascial trigger points in upper trapezius, subscapularis, anterior fibers of deltoid and supraspinatus muscle

Exclusion Criteria:

* Cervical Radiculopathies
* Thoracic outlet syndrome
* Rotator cuff tear
* Diabetes mellitus.
* Patients with any neurological disorder like hemiplegia.
* Fracture in and around shoulder

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-09-14 (Actual); Primary Completion 2023-04-02 (Actual); Study Completion 2023-04-02 (Actual)

PRIMARY OUTCOMES:
Numerical Rating Scale (NRS): | 4th week
  In a Numerical Rating Scale (NRS), patients are asked to circle the number between 0 and 10, 0 and 20 or 0 and 100 that fits best to their pain intensity [1]. Zero usually represents 'no pain at all' whereas the upper limit represents 'the worst pain ever possible.

SECONDARY OUTCOMES:
Range of motion | 4th week
  A goniometer is an instrument that measures the available range of motion at a joint. The art and science of measuring the joint ranges in each plane of the joint are called goniometry.
Shoulder Pain and Disability Index (SPADI): | 4th week
  The Shoulder Pain and Disability Index (SPADI) is a self-administered questionnaire that consists of two dimensions, one for pain and the other for functional activities. The pain dimension consists of five questions regarding the severity of an individual's pain. Functional activities are assessed with eight questions designed to measure the degree of difficulty an individual has with various activities of daily living that require upper-extremity use. The SPADI takes 5 to 10 minutes for a patient to complete and is the only reliable and valid region-specific measure for the shoulder.
  To answer the questions, patients place a mark on a 10cm visual analogue scale for each question. Verbal anchors for the pain dimension are 'no pain at all' and 'worst pain imaginable', and those for the functional activities are 'no difficulty' and 'so difficult it required help'. The scores from both dimensions are averaged to derive a total score.
Manual Muscle Testing (MMT): | 4th week
  Manual muscle testing (MMT) is a very common practice of orthopedic examination specifically designed to assess function and strength of various muscles, usually when rehabilitating sports injuries or recovering from an illness, MMT grades are usually labelled with the following terms: "zero," "trace," "poor," "fair," "good," and "normal." In addition, manual muscle testing grades can be further described using a numerical scale from 0 through 5.

CONTACTS AND LOCATIONS:
Overall Officials: KINZA ANWAR, MS-OMPT, Principal Investigator — RIPHAH INTERNATIONAL UNIVERSITY,ISLAMABAD,PAKISTAN
Locations (1):
- Bacha Khan Medical Complex Swabi (BKMCS) and District Headquarter Hospital (DHQ) Swabi., Swabi, Pakistan

IPD SHARING:
Plan to Share IPD: No